CLINICAL TRIAL: NCT07370987
Title: Prevention of Postoperative Pancreatic Fistula Following Pancreaticoduodenectomy by Preoperative Radiotherapy: a Phase 2 Trial
Brief Title: Prevention of Postoperative Pancreatic Fistula Following Pancreaticoduodenectomy by Preoperative Radiotherapy : a Phase 2 Trial
Acronym: PreFiR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP240932; IDRCB : 2025-A00206-43 (Other: ANSM)
Record Dates: First submitted 2025-09-09; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Fistula; Pancreaticoduodenectomy
Keywords: Pancreatic fistula; Surgery; pancreaticoduodenectomy; Radiotherapy
MeSH Terms: conditions — Pancreatic Fistula | interventions — Radiosurgery; Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Other): All patients enrolled in the trial and responding to inclusion/exclusion criteria will receive A dose of 20 Gy delivered in 2 fractions of 10 Gy, 1 day apart, of preoperative stereotactic radiotherapy targeting the isthmus of the pancreas over a 4 cm area that corresponds to the future anastomosis zone
  Interventions: Other: Stereotactic radiotherapy / pancreaticoduodenectomy

INTERVENTIONS:
Other: Stereotactic radiotherapy / pancreaticoduodenectomy — A dose of 20 Gy delivered in 2 fractions of 10 Gy, 1 day apart, of preoperative stereotactic radiotherapy Surgery : pancreaticoduodenectomy

SUMMARY:
Design of the study Prospective, single arm, multicentric, phase II open trial Number of participating sites 14 French centers of HPB Surgery departments associated with 14 Radiation Oncology Departments.

Implementation of the study A screening of eligible patients will be made locally by the referring surgeon of each centre based on patient medical records.

* Inclusion visit at the first surgical consultation (W-3 to D1) (V0) The inclusion visit will be done by the surgeon within 3 weeks before the first radiation oncologist visit
* D1 (V1): first radiation oncologist visit
* W2 (+/- 3D) and W4 (+/- 3D) (V2 et V3): Preoperative simulation process and treatment delivery
* A first visit at W+2 (+/- 3 D) will be mandatory to validate the positioning of the target volume by CBCT with IV constrast or MRI
* Then to start of the administration of radiotherapy at W+4 (+/- 3 D): Radiotherapy with 20 Gy, in 2 fraction of 10Gy with a one-day gap, so over a total period of 3

W9 ( +/- 1W) (V4): post-radiotherapy follow-up

- Preoperative visit Day-1 before PD (V5)

W10 (+/- 1W) (V6):

* Pancreaticoduodenectomy and post operative hospitalisation W14 (+/- 1W) (V7): follow up with surgeon (30 days after pancreaticoduodenectomy)
* W22 (+/-1W) (V8): follow up with surgeon (90 days after pancreaticoduodenectomy)
* W34 (+/-1W) (V9): Last study visit (radiation oncologist) (6 months after pancreaticoduodenectomy) Medical follow-up by radiation oncologist at 6 months after surgery to assess the occurrence of potential late toxicities due to radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 45 years old
* Candidate for pancreaticoduodenectomy by laparotomy
* Body mass index (BMI) ≥ 25kg/m2
* Diameter of main pancreatic duct (MPD) < 3 mm on preoperative CT scan or MRI at the isthmus of the pancreas (future pancreatic section area)
* Affiliation to a social security system (AME excepted)
* Signed informed consent

Exclusion Criteria:

* Surgery indication : Chronic pancreatitis
* Surgery indication : Pancreatic ductal adenocarcinoma
* History of syndromic or hereditary pancreatic tumor
* Contraindication to pancreaticoduodenectomy
* Planned multivisceral resection involving organs or parts of organs not normally involved in pancreatico-duodenectomy
* Planned external drainage of the main pancreatic duct at the end of the surgery
* Neoadjuvant treatment planned or performed by chemotherapy or radiotherapy
* History of chronic hepatitis (F3) or cirrhosis (F4)
* Contraindication to radiotherapy
* Previous history of abdominal radiotherapy
* Extended pancreatic resection on the left beyond the radiotherapy area (left of the pancreatic isthmus)
* History of complicated peptic ulcer
* Patient treated for less than 4 weeks for an ulcer
* History of pancreatic surgery
* Ongoing pregnancy (confirmed by a test beta-HCG) or breast feeding or absence of birth control
* Patients with a active pathology or history that may interfere with the study in progress or the interpretation of its results according to the investigator
* Patients with a history or suspicion of non-compliance with medical regimens or will be unable to complete the entire study
* Treatment with systemic corticosteroids (excluding inhaled corticosteroids)
* Participation in another interventional clinical study (RIPH1, clinical investigation or clinical trial) or exclusion period set after the study
* Protected persons under legal guardianship or conservatorship

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients at W22 (within 90 days from surgery) without grade B/C postoperative pancreatic fistula (POPF) | Week 22
  Postoperative fistula grade B and C is defined according to the last ISGPS classification of 2016 and will be adjudicated by independant experts.

SECONDARY OUTCOMES:
To assess overall surgical complication rate at W22 (90 days after surgery) | Week 22
  defined as a grade 1 to 5 according to the Dindo-Clavien classification complications occurring within 3 month from surgery
To assess severe surgical complication rate at W22 (90 days after surgery) | Week 22
  defined as a grade 3 to 5 according to the Dindo-Clavien classification complications occurring within 3 month from surgery
To assess, during surgery (W10), the hardness of pancreas texture on the specimen after resection with a durometer | Week 10
  determined intraoperatively by Durometer measurement of the radiated and irradiated pancreatic tissue in Shore OO
To assess, during surgery (W10), the hardness of pancreas texture on the specimen after resection by the surgeon | Week 10
  Determined intraoperatively by the pancreatic surgeon. Texture is scaled as soft/intermediate/hard at W10
To assess, during surgery (W10), technical difficulties added by radiotherapy, according to the surgeon | Day of surgery- Week 10
  Determined by 2 questions
  * To what extent was the surgery complicated by the radiotherapy? (Answers: 1 - not complicated; 2 - slightly complicated; 3 - clearly complicated; 4 - severely complicated; 5 - impossible)
  * Did you have to adapt the surgical plan due to the administration of radiotherapy? (Answers: Yes/No)
To assess on a pathological point of view the resected specimen at W14 | Day of surgery-week 14
  determined by the pathologist by evaluation of macroscopic differences between radiated and irradiated pancreatic tissue.
  - The extent and distribution of fibrosis and fat infiltration were evaluated using the score established by Rebours et al. in intra- and extralobular locations
To assess on a pathological point of view the resected specimen at W14 | Day of surgery-week 14
  determined by the pathologist by evaluation of macroscopic differences between radiated and irradiated pancreatic tissue.
  - Fibrosis quantification was also assessed by determining the area of collagen using Sirius red staining (as performed in FIBROPANC trial)
Pancreatic functionnal outcomes at W22 (de novo diabetes) | Week 22
  Determined by
  - De novo diabetes : In accordance with French and European recommendations, diabetes is diagnosed if fasting blood glucose is greater than or equal to 1.26 g/L on two occasions, or greater than or equal to 2 g/L at any time of the day, or if HbA1c is greater than 6.5%
Pancreatic functionnal outcomes at W22 (exocrine pancreatic insufficiency) | Week 22
  Determined by
  - Exocrine pancreatic insufficiency: A fecal elastase level < 100 mg/g stool is commonly accepted for diagnosing severe exocrine pancreatic insufficiency, a fecal elastase level between 100 and 200 mg/g indicates moderate exocrine pancreatic insufficiency, and a level > 200 mg/g stool rules out exocrine pancreatic insufficiency
To assess mortality rate at W22 | Week 22
To assess overall length of hospital stay after surgery | Up to Week 34
  Length of hospital stay between the operation and the day of discharge from hospital
To assess readmission rate at W22 | Week 22
  Proportion of readmission at W22, whatever the cause
To assess radiation-induced complications rate, overall and by grade at W9, W10, W14, W22, W34 | Week 9, Week 10, Week 14, Week 22 and Week 34
  to CTCAE classification (Common Terminology Criteria for Adverse Events), overall and by grade (grade 1 to 5)
To assess safety of radiotherapy at W9, and W34 | Week 9 and Week 34
  Proportion of patients at W9 and W34 who underwent at least one side effects of radiotherapy among gastritis or gastric bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Department of HPB Surgery, Hospital Pitié Salpétrière, Paris, France

IPD SHARING:
Plan to Share IPD: No